CLINICAL TRIAL: NCT06773442
Title: Assessment of Shoulder Rehabilitation Practices and Documentation Protocols at Rphah Rehabilitation Center, Lahore A Comprehensive Analysis
Brief Title: Assessment of Shoulder Rehabilitation Practices and Documentation Protocols at Riphah Rehabilitation Center
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/RCR&AHS24/37
Record Dates: First submitted 2024-07-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Pain; Shoulder Impingement; Rotator Cuff Injury
Keywords: shoulder pains; shoulder impingement; ,shoulder documentation
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP A:Rehabilitation Practices Group:: Objective: Evaluate the effectiveness and quality of shoulder rehabilitation practices.
  Data Collection, Observation of rehabilitation sessions: Record types of exercises, therapy techniques, patient engagement, and therapist-patient interactions.
  Interviews with rehabilitation professionals: Gather insights into their approaches, challenges faced, and perceived effectiveness of rehabilitation strategies.
  Analysis:
  Assess adherence to established rehabilitation protocols. Evaluate patient outcomes such as pain levels, range of motion, and functional status.
  Compare observed practices with evidence-based guidelines for shoulder rehabilitation.
  Findings:
  Identify strengths and weaknesses in current rehabilitation practices. Highlight areas where improvements or modifications may be necessary.
  Interventions: Other: Rehabilitation Practices Group
- GROUP B:Documentation Protocols Group: Objective: Assess the completeness, accuracy, and organization of documentation related to shoulder rehabilitation.
  Data Collection:
  Review of patient records and documentation: Evaluate the quality and consistency of documentation practices, including initial evaluations, progress notes, and discharge summaries.
  Interviews with rehabilitation staff: Collect feedback on documentation protocols, challenges encountered, and perceived adequacy of documentation practices.
  Analysis:
  Assess the clarity and comprehensiveness of documentation. Evaluate adherence to documentation protocols and standards. Identify any deficiencies or inconsistencies in documentation practices.
  Findings:
  Highlight strengths and weaknesses in current documentation protocols. Identify areas for improvement, such as standardizing documentation templates or providing training on effective documentation practices.
  Recommendations:
  Propose strategies to enhance documentation quality and consistency.
  Interventions: Other: Documentation Protocols Group

INTERVENTIONS:
Other: Rehabilitation Practices Group — Evidence-Based Training Program:Develop a structured training program for rehabilitation professionals focusing on evidence-based shoulder rehabilitation practices.
  Clinical Mentorship and Supervision:Implement a mentorship program where experienced rehabilitation professionals provide guidance and support to junior staff members.
  Standardization of Rehabilitation Protocols:Review and standardize rehabilitation protocols for common shoulder conditions based on current evidence and best practices.
  Patient-Centered Care Approach:Adopt a patient-centered approach to shoulder rehabilitation, emphasizing shared decision-making and individualized treatment plans Outcome Monitoring and Quality Improvement:Use standardized outcome measures to evaluate improvements in pain, function, range of motion, and patient satisfaction.
  Groups: GROUP A:Rehabilitation Practices Group:
Other: Documentation Protocols Group — Training and Education Program:Develop and implement a training program for rehabilitation professionals aimed at enhancing their knowledge and skills in shoulder rehabilitation practices and documentation protocols.
  Standardization of Protocols:Review and update existing rehabilitation protocols to ensure alignment with current evidence-based guidelines and best practices.
  Quality Assurance Measures:Establish a system for ongoing monitoring and evaluation of shoulder rehabilitation practices and documentation protocols.
  Patient Education and Engagement:Develop educational materials and resources for patients undergoing shoulder rehabilitation to enhance their understanding of treatment goals, exercises, and self-management strategies.
  Outcome Monitoring and Evaluation:Implement a system for monitoring and evaluating patient outcomes, including pain levels, range of motion, functional status, and satisfaction with rehabilitation services.
  Groups: GROUP B:Documentation Protocols Group

SUMMARY:
This study aims to evaluate Riphah Rehabilitation Center's shoulder rehabilitation procedures and documentation guidelines. The study will specifically assess the efficacy of shoulder rehabilitation procedures, their methodology, and the techniques employed to record patient improvement. In order to make sure the centre adheres to best practices, improves patient care, and keeps accurate records for better treatment outcomes, the study intends to identify areas of strength and potential improvements in both the rehabilitation techniques and documentation processes. The evaluation's findings will improve the center's operational effectiveness and clinical practices.

Target Audience:Healthcare Professionals (such as physicians, physiotherapists, and rehabilitation therapists): This study will assist guide evidence-based strategies for managing shoulder injuries and offer insights into contemporary rehabilitation procedures.

Centre Administration: For better patient care, resource management, and operational efficiency, the results will point out areas where documentation and treatment protocols should be strengthened.

Patients and Families: In the end, the study will improve rehabilitation results, increasing the likelihood that patients will heal from shoulder injuries more quickly and completely.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing shoulder rehabilitation at Rphah Rehabilitation Center.
* Rehabilitation protocols implemented within the center.
* Documented cases with sufficient information for analysis.
* Both acute and chronic shoulder conditions

Exclusion Criteria:

* Patients with shoulder conditions not requiring rehabilitation.
* Cases lacking adequate documentation.
* Rehabilitation protocols not specific to shoulder conditions.
* Patients with comorbidities significantly affecting rehabilitation outcomes.

Ages: 23 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients Undergoing Shoulder Rehabilitation:
  Include patients who have undergone or are currently undergoing rehabilitation specifically for shoulder injuries, conditions, or surgeries.
  Consider both inpatients and outpatients receiving rehabilitation services at Rphah Rehabilitation Center.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-26 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity During Shoulder Rehabilitation Treatment | Baseline and 4 weeks (post-intervention)
  Pain severity will be assessed using a Numerical Rating Scale (0-10), where 0 indicates no pain and 10 indicates the worst imaginable pain. Both groups will receive 2 treatment sessions per week. Pain assessments will be made at baseline (pre-intervention) and at the end of the 4-week intervention (post-intervention) to evaluate changes in pain severity.
  Measurement Unit: Numerical Rating Scale (0-10), where 0 = no pain, 10 = worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hashim, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah Rehabilitation Center, Lahore, Punjab Province
  - Riphah Rehabilitation Center, Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith BA, Fields CJ, Fernandez N. Physical therapists make accurate and appropriate discharge recommendations for patients who are acutely ill. Phys Ther. 2010 May;90(5):693-703. doi: 10.2522/ptj.20090164. Epub 2010 Mar 18. PMID 20299410
- [Background] Scalzitti DA. On
- [Background] De Villers MJ. Documentation of preventive education and screening for osteoporosis. Outcomes Manag. 2003 Jan-Mar;7(1):28-32. PMID 12593123
- [Background] Ajami S, Arab-Chadegani R. Barriers to implement Electronic Health Records (EHRs). Mater Sociomed. 2013;25(3):213-5. doi: 10.5455/msm.2013.25.213-215. PMID 24167440